CLINICAL TRIAL: NCT06394089
Title: Effect of Degenerative Spondylolisthesis on the Clinical Outcome of Unilateral Biportal Endoscopy for Lumbar Spinal Stenosis: a Single-center, Prospective Cohort Trial Protocol
Brief Title: Effect of Degenerative Spondylolisthesis on the Clinical Outcome of Unilateral Biportal Endoscopy for Lumbar Spinal Stenosis: Study Protocol
Status: Recruiting | Type: Observational
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-P2-293-01
Record Dates: First submitted 2024-04-07; First posted 2024-05-01 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Degenerative Spondylolisthesis; Lumbar Spinal Stenosis
MeSH Terms: conditions — Spinal Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (2):
- DS Group: Patients with degenerative spondylolisthesis Meyerding grade Ⅰ (slippage >3 mm but <25%) will be identified as having lumbar spinal stenosis combined with degenerative spondylolisthesis and will be allocated to the DS group.
- Non-DS Group: Patients not with degenerative spondylolisthesis will be identified as having lumbar spinal stenosis only and will be allocated to the Non-DS group.

SUMMARY:
A single-center, prospective cohort trial aims to provide stronger evidence regarding the impact of degenerative spondylolisthesis on the clinical outcome of unilateral biportal endoscopy for lumbar spinal stenosis

ELIGIBILITY:
Inclusion Criteria:

* Age range: 50-80 years
* Diagnosis of LSS affecting 1-2 vertebral levels
* Predominant manifestation of neurogenic intermittent claudication, with ineffective conservative treatment for at least 3 months
* Presence of lumbar DS of less than grade II and absence of spine instability
* Willingness to participate in the study and complete follow-up assessments.

Exclusion Criteria:

* Diagnosis of isthmic lumbar spondylolisthesis or lumbar DS of grade ≥II
* Evidence of instability at the affected vertebral level (intervertebral angle change > 15° and/or vertebral translation ≥ 4.5 mm in standing flexion-extension radiographs of the lumbar spine)
* History of prior surgery at the affected vertebral level
* Presence of scoliosis with a Cobb angle >20º
* Presence of other conditions affecting the lumbar spine (infection, tumor, fracture, neurological diseases, and others)
* Medical disorders that preclude surgical tolerance
* Participation in other clinical research projects related to the treatment of lumbar spinal stenosis.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible patients with LSS who are scheduled to undergo UBE-based decompression, performed by an experienced spine surgeon at Beijing Friendship Hospital, will be recruited from the outpatient clinic for this study.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Oswestry Disability Index (ODI) | From enrollment to the end of follow-up at 2 year
  0-100%, the higher the score, the more severe the lumbar spine dysfunction

SECONDARY OUTCOMES:
X-ray | From enrollment to the end of follow-up at 2 year
  Progression of lumbar spondylolisthesis, assessed by postoperative lumbar radiography; (2) Measurement of sagittal translation, segmental angulation, and posterior opening based on postoperative standing flexion-extension radiographs
Computed tomography (CT) scan | From enrollment to the end of follow-up at 2 year
  Assessment of bone resection area and preservation rate of the facet joint using postoperative computed tomography (CT) scans
Magnetic resonance imaging (MRI) | From enrollment to the end of follow-up at 2 year
  Calculation of the enlargement ratio of the dural sac based on postoperative magnetic resonance imaging (MRI)
Surgical complication | From enrollment to the end of follow-up at 2 year
  Any adverse events will be recorded to evaluate the safety of decompression using UBE for LSS with or without DS
Visual analog scale (VAS) score for lower back pain | From enrollment to the end of follow-up at 2 year
  0-10, the higher the score, the more severe the pain
Visual analog scale (VAS) score for leg pain | From enrollment to the end of follow-up at 2 year
  0-10, the higher the score, the more severe the pain
Operative time | Immediately after the surgery
  Time to perform the operation
Intraoperative blood loss | Immediately after the surgery
  B、 Blood loss during the surgery
Postoperative hospital stays | Immediately after the discharge
  Number of days in hospital after operation
Japanese Orthopaedic Association (JOA) score | From enrollment to the end of follow-up at 2 year
  0-29, the higher the score, the better the lumbar spine function
Modified MacNab criteria | From enrollment to the end of follow-up at 2 year
  According to satisfaction, it is divided into four levels: excellent, good, acceptable, and poorexcellent, good, fair, and poor
Improvement ratio of Visual analog scale (VAS) score for lower back pain | From enrollment to the end of follow-up at 2 year
  Improvement ratio= (preoperative VAS-postoperative VAS/preoperative VAS, ranging from 0-100%, the higher the score, the better the improment of symptoms
Improvement ratio of Visual analog scale (VAS) score for leg pain | From enrollment to the end of follow-up at 2 year
  Improvement ratio= (preoperative VAS-postoperative VAS/preoperative VAS, ranging from 0-100%, the higher the score, the better the improment of symptoms
Improvement ratio of Japanese Orthopaedic Association (JOA) score | From enrollment to the end of follow-up at 2 year
  Improvement ratio= (postoperative JOA-preoperative JOA/preoperative VAS, ranging from 0-100%, the higher the score, the better the improment of spinal function
Improvement ratio of Oswestry Disability Index (ODI) | From enrollment to the end of follow-up at 2 year
  Improvement ratio= (preoperative ODI-postoperative ODI)/preoperative ODI, ranging from 0-100%, the higher the score, the better the improment of symptoms
White blood cell count | From enrollment to 3 days after surgery
  White blood cell count of venous blood
Percentage of neutrophils (N%) | From enrollment to 3 days after surgery
  The proportion of neutrophils relative to the total white blood cell count
C-reactive protein level | From enrollment to 3 days after surgery
  The level of C-reactive protein in blood
Creatine kinase level | From enrollment to 3 days after surgery
  The level of creatine kinase in blood
Lactate dehydrogenase level | From enrollment to 3 days after surgery
  The level of Lactate dehydrogenase in blood
Myoglobin level | From enrollment to 3 days after surgery
  The level of myoglobin in blood

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Friendship Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liu Y, Li G, Yu L, Sun H, Zhu B, Fei Q, Lo Y, Yang Y, Tan H, Li X. Degenerative spondylolisthesis and unilateral biportal endoscopic decompression for lumbar spinal stenosis: a single-center, prospective cohort trial protocol. BMC Musculoskelet Disord. 2025 Oct 1;26(1):900. doi: 10.1186/s12891-025-09179-6. PMID 41034885